CLINICAL TRIAL: NCT04595253
Title: Professor, School of Nursing, China Medical University Hospital, Principal Investigator
Brief Title: The Effectiveness of Acupressure for Managing Postoperative Pain and Anxiety in Patients With Thoracoscopic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wei-Fen Ma (Other)
Collaborators: China Medical University Hospital (Other)
Responsible Party: Sponsor-Investigator, Wei-Fen Ma, Professor, School of Nursing, China Medical University Hospital
Organization: China Medical University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CMUH109-REC2-131
Record Dates: First submitted 2020-10-09; First posted 2020-10-20 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Lung Diseases
Keywords: acupressure; thoracoscopic surgery; acute pain; anxiety; comfort
MeSH Terms: conditions — Lung Diseases; Acute Pain; Anxiety Disorders | interventions — Acupressure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- acupressure (Experimental): After recruitment, participants will be randomized to receive acupressure or control group. In the acupressure group, participants will receive acupressure treatment.
  Interventions: Other: acupressure
- routine care (No Intervention): After recruitment, participants will be randomized to receive acupressure or control group. In the control group, participants will receive routine care, including routine pain control.

INTERVENTIONS:
Other: acupressure — The acupressure involves the " Vaccaria Semen" within skin-colored adhesive tape that placed on the "Neiguan" and "Shenmen" acupoints as an intervention measure. Continue to massage the acupoints with fingertips for 10 minutes, 3 times per day (8 and 12 in the morning, and 4 in the afternoon) . The adhesive tape will be retained in situ for 2 days.
  Arms: acupressure

SUMMARY:
The purpose of this study is to explore the effectiveness of acupressure for managing postoperative pain, anxiety, analgesia consumption, early ambulation, and comfort in patients with thoracoscopic surgery.

DETAILED DESCRIPTION:
Thoracoscopic surgery is the surgical used to removal of a section or a segment of a lung lobe. One US national survey reported that 80% of patients undergoing pulmonary surgery experienced acute pain. 75-86% of these patients pointed out that experienced moderate, severe, or extreme pain, especially, on the 1st day after thoracoscopic surgery. However, inappropriate pain management after surgery is associated with limited the healing process, increased workload of heart, prolonged pulmonary rehabilitation, and increased medical costs, and can be a prediction of developing chronic pain. Acupressure is a nonpharmacological treatment for the management of postoperative pain. Recent studies have found that the application of acupressure is effective in decreasing operative pain intensity, morphine related side effects, and opioid consumptions after surgery. However, there was no further research about the role of acupressure applied to thoracoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* pulmonary lung disease and will be scheduled to undergo a thoracoscopic wedge resection, segmentectomy, or lobectomy.
* American Society of Anesthesiologist physical status of Classes I-II,
* both forearms without missing limbs or arteriovenous fistula
* ability to communicate in Taiwanese or Chinese, and
* agreement to participate in this study.

Exclusion Criteria:

* diagnosed as malignant neoplasm with lung meta,
* Had a stroke or peripheral vascular disease
* Platelet count less than 20 x 10^3/mm^3
* Using the patient controlled analgesia, and
* any known mental illness or memory dysfunction.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-09-20 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Pain:Changes from baseline pain scale at post-operative day 2, after intervention. | Measure at before operation day, 7 post meridiem (PM), before operation; post-operative day1, 8 ante meridiem (AM), before intervention; post-operative day 1, 5 PM, after intervention; and post-operative day 2, 5 PM, after intervention
  as assessed by Visual Analogue Scale-Pain (VAS-P). The VAS-P scale is comprised of a horizontal line 100mm long with the indication "no pain" to the left and "worst possible pain" to the right. possible scores varied between 0-100. A higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Anxiety | Measure at before operation day, 7 post meridiem (PM), before operation; post-operative day1, 9 ante meridiem (AM), before intervention; post-operative day 1, 5 PM, after intervention; and post-operative day 2, 5 PM, after intervention.
  as assessed by Visual Analogue Scale-Anxiety(VAS-A). The VAS-A scale is comprised of a horizontal line 100mm long with the indication "no anxiety" to the left and "worst possible anxiety" to the right. possible scores varied between 0-100. A higher scores mean a worse outcome.
Anxiety | Time Frame: Measure at before operation day, 7 post meridiem (PM), before operation; post-operative day1, 8 ante meridiem (AM), before intervention; and post-operative day 2, post meridiem (PM), after intervention.
  as assessed by State-Trait Anxiety Inventory (STAI) Y form (STAI-Y1). It is 20 questions, which were rated from 1-4. Possible scores varied between 20-80. A STAI-Y1 score>40 as evidence of a state of anxiety.

OTHER OUTCOMES:
Analgesia Consumption | during the whole admission, an average of 4 day.
  Injection time of morphine and ketorolac would be recorded.
Comfort | Measure at before operation day,7 post meridiem (PM), before operation; post-operative day 1, 8 ante meridiem (AM), before intervention; and post-operative day 2, 5pm, after intervention
  as assessed by Shortened General Comfort Questionnaire
Heart rate variability | Measure at before operation day, 7 post meridiem (PM), before operation; post-operative day1, 8 ante meridiem (PM), before intervention; post-operative day 1, 5 post meridiem (PM), after intervention; and post-operative day 2, 5 PM, after intervention.
  as assessed by Nexus-10, wireless Biofeedback/Neurofeedback system
Early ambulation | The first ambulation time after operation would be recorded, assessed up to 7 days.
  The first ambulation time: act to walk with or without any kind of assistant after operation.

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Fen Ma, Ph.D, Principal Investigator — China Medical University, China
Locations (1):
- China Medical University, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amico, T. A. D. (2007). Thoracoscopic Lobectomy. Journal of Medical Sciences, 27(3), 95-100. https://doi.org/10.6136/JMS.2007.27(3).095
- [Background] Apfelbaum JL, Chen C, Mehta SS, Gan TJ. Postoperative pain experience: results from a national survey suggest postoperative pain continues to be undermanaged. Anesth Analg. 2003 Aug;97(2):534-540. doi: 10.1213/01.ANE.0000068822.10113.9E. PMID 12873949
- [Background] Au DW, Tsang HW, Ling PP, Leung CH, Ip PK, Cheung WM. Effects of acupressure on anxiety: a systematic review and meta-analysis. Acupunct Med. 2015 Oct;33(5):353-9. doi: 10.1136/acupmed-2014-010720. Epub 2015 May 22. PMID 26002571
- [Background] Batvani M, Yousefi H, Valiani M, Shahabi J, Mardanparvar H. The Effect of Acupressure on Physiological Parameters of Myocardial Infarction Patients: A Randomized Clinical Trial. Iran J Nurs Midwifery Res. 2018 Mar-Apr;23(2):143-148. doi: 10.4103/ijnmr.IJNMR_83_16. PMID 29628963
- [Background] Boker A, Brownell L, Donen N. The Amsterdam preoperative anxiety and information scale provides a simple and reliable measure of preoperative anxiety. Can J Anaesth. 2002 Oct;49(8):792-8. doi: 10.1007/BF03017410. PMID 12374706
- [Background] Chang LH, Hsu CH, Jong GP, Ho S, Tsay SL, Lin KC. Auricular acupressure for managing postoperative pain and knee motion in patients with total knee replacement: a randomized sham control study. Evid Based Complement Alternat Med. 2012;2012:528452. doi: 10.1155/2012/528452. Epub 2012 Jul 10. PMID 22844334
- [Background] Chang S. The meridian system and mechanism of acupuncture: a comparative review. Part 3: Mechanisms of acupuncture therapies. Taiwan J Obstet Gynecol. 2013 Jun;52(2):171-84. doi: 10.1016/j.tjog.2013.04.005. PMID 23915848
- [Background] Chang S. The meridian system and mechanism of acupuncture-a comparative review. Part 1: the meridian system. Taiwan J Obstet Gynecol. 2012 Dec;51(4):506-14. doi: 10.1016/j.tjog.2012.09.004. PMID 23276552
- [Background] Chen JS, Cheng YJ, Hung MH, Tseng YD, Chen KC, Lee YC. Nonintubated thoracoscopic lobectomy for lung cancer. Ann Surg. 2011 Dec;254(6):1038-43. doi: 10.1097/SLA.0b013e31822ed19b. PMID 21869676
- [Background] Chen T, Wang K, Xu J, Ma W, Zhou J. Electroacupuncture Reduces Postoperative Pain and Analgesic Consumption in Patients Undergoing Thoracic Surgery: A Randomized Study. Evid Based Complement Alternat Med. 2016;2016:2126416. doi: 10.1155/2016/2126416. Epub 2016 Mar 17. PMID 27073400
- [Background] Coutaux A. Non-pharmacological treatments for pain relief: TENS and acupuncture. Joint Bone Spine. 2017 Dec;84(6):657-661. doi: 10.1016/j.jbspin.2017.02.005. Epub 2017 Feb 20. PMID 28219657
- [Background] Danoff JR, Goel R, Sutton R, Maltenfort MG, Austin MS. How Much Pain Is Significant? Defining the Minimal Clinically Important Difference for the Visual Analog Scale for Pain After Total Joint Arthroplasty. J Arthroplasty. 2018 Jul;33(7S):S71-S75.e2. doi: 10.1016/j.arth.2018.02.029. Epub 2018 Feb 22. PMID 29567002
- [Background] Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. No abstract available. PMID 8598068
- [Background] Endler NS, Kocovski NL. State and trait anxiety revisited. J Anxiety Disord. 2001 May-Jun;15(3):231-45. doi: 10.1016/s0887-6185(01)00060-3. PMID 11442141
- [Background] Engen DJ, Carns PE, Allen MS, Bauer BA, Loehrer LL, Cha SS, Chartrand CM, Eggler EJ, Cutshall SM, Wahner-Roedler DL. Evaluating efficacy and feasibility of transcutaneous electrical nerve stimulation for postoperative pain after video-assisted thoracoscopic surgery: A randomized pilot trial. Complement Ther Clin Pract. 2016 May;23:141-8. doi: 10.1016/j.ctcp.2015.04.002. Epub 2015 Apr 20. PMID 25935320
- [Background] Erdogan M, Erdogan A, Erbil N, Karakaya HK, Demircan A. Prospective, Randomized, Placebo-controlled Study of the Effect of TENS on postthoracotomy pain and pulmonary function. World J Surg. 2005 Dec;29(12):1563-70. doi: 10.1007/s00268-005-7934-6. PMID 16331341
- [Background] Fletcher D, Martinez V. Opioid-induced hyperalgesia in patients after surgery: a systematic review and a meta-analysis. Br J Anaesth. 2014 Jun;112(6):991-1004. doi: 10.1093/bja/aeu137. PMID 24829420
- [Background] Frödin, M., & Warrén Stomberg, M. (2014). Pain management after lung surgery. Nursing Reports, 4(1). https://doi.org/10.4081/nursrep.2014.3225
- [Background] Fu, J., & Yang, M. (2019). The Yellow Emperor's Classic of Medicine - Essential Questions: Translation of Huangdi Neijing Suwen. WORLD SCIENTIFIC. https://doi.org/10.1142/11080
- [Background] Gan TJ. Poorly controlled postoperative pain: prevalence, consequences, and prevention. J Pain Res. 2017 Sep 25;10:2287-2298. doi: 10.2147/JPR.S144066. eCollection 2017. PMID 29026331
- [Background] Gan TJ, Habib AS, Miller TE, White W, Apfelbaum JL. Incidence, patient satisfaction, and perceptions of post-surgical pain: results from a US national survey. Curr Med Res Opin. 2014 Jan;30(1):149-60. doi: 10.1185/03007995.2013.860019. Epub 2013 Nov 15. PMID 24237004
- [Background] Gupta A, Kaur K, Sharma S, Goyal S, Arora S, Murthy RS. Clinical aspects of acute post-operative pain management & its assessment. J Adv Pharm Technol Res. 2010 Apr;1(2):97-108. PMID 22247838
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Background] Hornblow AR, Kidson MA. The visual analogue scale for anxiety: a validation study. Aust N Z J Psychiatry. 1976 Dec;10(4):339-41. doi: 10.3109/00048677609159523. No abstract available. PMID 1071419
- [Background] Hsiung DY, Liu CW, Cheng PC, Ma WF. Using non-invasive assessment methods to predict the risk of metabolic syndrome. Appl Nurs Res. 2015 May;28(2):72-7. doi: 10.1016/j.apnr.2014.12.001. Epub 2014 Dec 17. PMID 25908541
- [Background] Huskisson EC. Measurement of pain. Lancet. 1974 Nov 9;2(7889):1127-31. doi: 10.1016/s0140-6736(74)90884-8. No abstract available. PMID 4139420
- [Background] Kaplowitz J, Papadakos PJ. Acute pain management for video-assisted thoracoscopic surgery: an update. J Cardiothorac Vasc Anesth. 2012 Apr;26(2):312-21. doi: 10.1053/j.jvca.2011.04.010. Epub 2011 Jun 25. No abstract available. PMID 21705236
- [Background] Kibler VA, Hayes RM, Johnson DE, Anderson LW, Just SL, Wells NL. Cultivating quality: early postoperative ambulation: back to basics. Am J Nurs. 2012 Apr;112(4):63-9. doi: 10.1097/01.NAJ.0000413460.45487.ea. No abstract available. PMID 22456575
- [Background] Kindler CH, Harms C, Amsler F, Ihde-Scholl T, Scheidegger D. The visual analog scale allows effective measurement of preoperative anxiety and detection of patients' anesthetic concerns. Anesth Analg. 2000 Mar;90(3):706-12. doi: 10.1097/00000539-200003000-00036. PMID 10702461
- [Background] Kolcaba K, Schirm V, Steiner R. Effects of hand massage on comfort of nursing home residents. Geriatr Nurs. 2006 Mar-Apr;27(2):85-91. doi: 10.1016/j.gerinurse.2006.02.006. PMID 16638478
- [Background] Kuroda H, Mizuno H, Dejima H, Watanabe K, Yoshida T, Naito Y, Sakao Y. A retrospective study on analgesic requirements for thoracoscopic surgery postoperative pain. J Pain Res. 2017 Nov 15;10:2643-2648. doi: 10.2147/JPR.S147691. eCollection 2017. PMID 29180890
- [Background] Ma WF, Liu YC, Chen YF, Lane HY, Lai TJ, Huang LC. Evaluation of psychometric properties of the Chinese Mandarin version State-Trait Anxiety Inventory Y form in Taiwanese outpatients with anxiety disorders. J Psychiatr Ment Health Nurs. 2013 Aug;20(6):499-507. doi: 10.1111/j.1365-2850.2012.01945.x. Epub 2012 Jul 5. PMID 22762356
- [Background] Mehta P, Dhapte V, Kadam S, Dhapte V. Contemporary acupressure therapy: Adroit cure for painless recovery of therapeutic ailments. J Tradit Complement Med. 2016 Jul 22;7(2):251-263. doi: 10.1016/j.jtcme.2016.06.004. eCollection 2017 Apr. PMID 28417094
- [Background] Nomori H, Horio H, Naruke T, Suemasu K. What is the advantage of a thoracoscopic lobectomy over a limited thoracotomy procedure for lung cancer surgery? Ann Thorac Surg. 2001 Sep;72(3):879-84. doi: 10.1016/s0003-4975(01)02891-0. PMID 11565674
- [Background] Pogatzki-Zahn EM, Segelcke D, Schug SA. Postoperative pain-from mechanisms to treatment. Pain Rep. 2017 Mar 15;2(2):e588. doi: 10.1097/PR9.0000000000000588. eCollection 2017 Mar. PMID 29392204
- [Background] Sharifi Rizi M, Shamsalinia A, Ghaffari F, Keyhanian S, Naderi Nabi B. The effect of acupressure on pain, anxiety, and the physiological indexes of patients with cancer undergoing bone marrow biopsy. Complement Ther Clin Pract. 2017 Nov;29:136-141. doi: 10.1016/j.ctcp.2017.09.002. Epub 2017 Sep 5. PMID 29122251
- [Background] Tamura M, Shimizu Y, Hashizume Y. Pain following thoracoscopic surgery: retrospective analysis between single-incision and three-port video-assisted thoracoscopic surgery. J Cardiothorac Surg. 2013 Jun 12;8:153. doi: 10.1186/1749-8090-8-153. PMID 23759173
- [Background] Wang Y, Tang H, Guo Q, Liu J, Liu X, Luo J, Yang W. Effects of Intravenous Patient-Controlled Sufentanil Analgesia and Music Therapy on Pain and Hemodynamics After Surgery for Lung Cancer: A Randomized Parallel Study. J Altern Complement Med. 2015 Nov;21(11):667-72. doi: 10.1089/acm.2014.0310. Epub 2015 Sep 2. PMID 26331434
- [Background] You WY, Yeh TP, Lee KC, Ma WF. A Preliminary Study of the Comfort in Patients with Leukemia Staying in a Positive Pressure Isolation Room. Int J Environ Res Public Health. 2020 May 22;17(10):3655. doi: 10.3390/ijerph17103655. PMID 32456113
- [Background] Wu CL, Raja SN. Treatment of acute postoperative pain. Lancet. 2011 Jun 25;377(9784):2215-25. doi: 10.1016/S0140-6736(11)60245-6. PMID 21704871
- [Background] World Health Organization. (1991). A Proposed Standard International Acupuncture Nomenclature: Report of a WHO Scientific Group. Annals of Internal Medicine, 115(4), 335. https://doi.org/10.7326/0003-4819-115-4-335_2
- [Result] Abouarab AA, Rahouma M, Kamel M, Ghaly G, Mohamed A. Single Versus Multi-Incisional Video-Assisted Thoracic Surgery: A Systematic Review and Meta-analysis. J Laparoendosc Adv Surg Tech A. 2018 Feb;28(2):174-185. doi: 10.1089/lap.2017.0446. Epub 2017 Nov 6. PMID 29106318
- See also: American Society of Anesthesiologists Physical Status Classification System. — https://www.asahq.org/standards-and-guidelines/asa-physical-status-classification-system

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-19): https://cdn.clinicaltrials.gov/large-docs/53/NCT04595253/Prot_SAP_000.pdf